#### MEDICAL RECORD

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

Date posted to web: 10/23/20

INSTITUTE: National Cancer Institute

STUDY NUMBER: 16-C-0048 PRINCIPAL INVESTIGATOR: Ravi Madan, M.D.

STUDY TITLE: Docetaxel and PROSTVAC for Metastatic Castration Sensitive Prostate Cancer

Continuing Review Approved by the IRB on 10/15/20 Amendment Approved by the IRB on 08/17/18 (H)

Standard

## INTRODUCTION

We invite you to take part in a research study at the National Institutes of Health (NIH).

First, we want you to know that:

Taking part in NIH research is entirely voluntary.

You may choose not to take part, or you may withdraw from the study at any time. In either case, you will not lose any benefits to which you are otherwise entitled. However, to receive care at the NIH, you must be taking part in a study or be under evaluation for study participation.

You may receive no benefit from taking part. The research may give us knowledge that may help people in the future.

Second, some people have personal, religious or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). If you have such beliefs, please discuss them with your NIH doctors or research team before you agree to the study.

Now we will describe this research study. Before you decide to take part, please take as much time as you need to ask any questions and discuss this study with anyone at NIH, or with family, friends or your personal physician or other health professional.

#### Why are you being asked to take part in this study?

You have been asked to take part in this research study because you have metastatic castrate-sensitive prostate cancer. Metastatic means your prostate cancer has spread outside of the areas around your prostate (usually the bones or other organs). Castrate-sensitive means your cancer can still be controlled by lowering the amount of testosterone in your body. This type of treatment is called androgen deprivation therapy (ADT) and it is one type of standard option. ADT treatment is not experimental. Your doctors will describe your treatment plan to you in detail before asking

PATIENT IDENTIFICATION

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or

• Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099

| Study | MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|---|
|---|---|---|

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

you to sign this consent form. You may be asked to sign a separate consent form for any treatment procedures not outlined in this consent.

### Why is this study being done?

Recently a clinical study showed that adding chemotherapy (docetaxel) for six infusions significantly extended the lives of men compared to those who were only treated with ADT alone. This study is being done to determine if combining a vaccine called PROSTVAC and the chemotherapy docetaxel along with androgen deprivation therapy (ADT) will work better.

Clinical work with PROSTVAC is based on the idea that the immune system (group of cells and organs in the body that recognize and fight infection) can be taught to find and kill certain cancer cells, in this case prostate cancer cells. This is a new vaccine treatment, which means that it is not approved for use on the general public and can only be used in a research study. In September of 2017, it was reported that a large (phase III) study of PROSTVAC alone did not show that this treatment could improve survival in advanced prostate cancer. (A phase III study is designed to lead to FDA approval and standard use of a therapy if the findings are positive.) The preliminary findings of the study suggest that PROSTVAC alone did not have an impact (positive or negative) on overall survival of patients treated. All patients had a similar length of survival regardless of treatment with vaccine alone or no treatment. However, the scientific reasoning to combine PROSTVAC with standard use docetaxel remains sound, and this study will continue. Furthermore, at this point neither this trial nor the phase III trial have suggested a safety concern for PROSTVAC.

In this study, you will be assigned to Arm C if you are a patient who has not started ADT or a patient who has started on ADT within the last 28 days. Otherwise, your treatment group (Arm A or Arm B) will be decided by a randomization process (chosen as if by the flip of a coin). Random assignment will be done with the help of a computer and you will be told on the day you start about your assigned group. You have an equal chance of being randomized to any of the two groups.. If you are randomized to Arm A, you will receive ADT for at least 28 days followed by docetaxel and then a vaccine called PROSTVAC. If you are in Arm B, you will receive ADT for at least 28 days followed by PROSTVAC and docetaxel, given 20-48 hours apart. If you are in Arm C, you will receive ADT for less than or equal to 28 days followed by PROSTVAC. After the vaccine treatment course is complete, the docetaxel course will be begin within 28 days of the last vaccine given.

It is important to note that in the clinical study that showed chemotherapy with ADT improved survival, the greatest benefit was seen in men with high volume disease (disease in more than 4 spots in the bones, including areas beyond the spine and pelvis, or disease in an organ). For patients with low volume disease (less than 4 areas in the bones, not beyond the ribs or pelvis, or not in an organ) the data is less clear. It appears with longer follow up there may not be a clear benefit of the chemotherapy in terms of overall survival (based on new data presented in the Fall

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

of 2016). Statistically speaking, this is not a perfect analysis and thus questions remain. Nonetheless, this treatment seems to be an appropriate option for "low volume" patients since patients with low volume of disease were eligible for the study which showed a benefit overall. Also, the treatment is well tolerated because more than 86% of the patients who started chemotherapy received all 6 infusions. The primary investigator or an associate investigator will discuss specifically how your disease relates to the data that is available. We also encourage you to discuss enrollment in this clinical trial with your primary oncologist to get a second opinion. For Arm C participants, chemotherapy will begin within 4 months of starting ADT and possibly sooner, depending on your disease. This trial was designed to remain consistent with the data this study is based on.

## How many people will take part in this study?

We plan to enroll up to 74 patients in the study.

#### **Description of Research Study**

#### What will happen if you take part in this research study?

#### Before you begin the study

You will need to have a physical exam, blood tests and scans to find out if you can be in the study. The exams and tests are part of regular cancer care and may be done even if you do not join the study. However, there are some extra exams, tests and procedures that you will need to have if you take part in this study. If you had some of the tests recently, they may not need to be repeated. The following is a list of what we need to make sure you can do this study:

- Medical history and physical exam.
- Blood tests including a complete blood count, chemistry panel, and prostate-specific antigen (PSA) levels.
- Electrocardiogram (ECG)
- Scans or other imaging studies
- Human immunodeficiency virus (HIV) test. HIV infection may disqualify you from this study. If you test positive for HIV, we will tell you what the results mean, how to find care, how to avoid infecting others, how we report newly diagnosed HIV infection.
- Hepatitis B and C. If these tests are positive, you will not be eligible to participate in the study because there is a possibility the vaccine may harm you.

Altogether, these tests will require about 100 ml (6 to 7 tablespoons) of blood.

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

## **During the study**

Once you agree to participate in this study and you are fit to join, you will be randomized to Arm A or Arm B or assigned to Arm C based on when you started ADT (Arm C will not be part of a randomization because it was added to the study after Arms A and B were nearly completed):

## • Arm A: ADT followed by docetaxel, then PROSTVAC

About 1-4 months after starting ADT, you will be given docetaxel by vein every three weeks for a total of six cycles. Docetaxel is a 1-hour infusion and patients are asked to take steroid pills by mouth or given steroids by vein before it is given to prevent side effects or allergic reactions. Docetaxel will be given on weeks 1,4,7,10,13, and 16. Three weeks after the last docetaxel infusion, you will be given the first vaccine injection called vaccinia-PROSTVAC (week 19). Two weeks after the first vaccine injection you will be given a booster injection called fowlpox-PROSTVAC. The first booster injection is given on week 21 and every 3 weeks for a total of 6 booster injections. Fowlpox-PROSTVAC will be given in weeks 21, 24, 27, 30, 33, and 36.

## • Arm B: ADT followed by docetaxel + PROSTVAC (given around the same time)

About 1-4 months after starting ADT, you will be given the first vaccine injection called vaccinia-PROSTVAC. Two weeks later you will be given a booster injection called fowlpox-PROSTVAC. Docetaxel is given by vein 20-48 hours after the booster injections. Docetaxel is a 1-hour infusion and patients are asked to take steroid pills by mouth or given steroids by vein before it is given to prevent side effects or allergic reactions. Docetaxel and fowlpox-PROSTVAC is given every 3 weeks for a total of six cycles. They will be administered on weeks 1,4,7,10,13, and 16.

# • ARM C: ADT followed by PROSTVAC, then Docetaxel (for patients who have not started ADT or who have been on ADT for less than 28 days)

Within 28 days of starting ADT you will be given vaccinia-PROSTVAC. This will be followed by 3-5 booster injections called fowlpox-PROSTVAC. The number of booster treatments you receive will be based on your disease and discussions between you and your doctor. Docetaxel will be initiated within 28 days of your last vaccine booster as discussed with your doctor, but not beyond 134 days (about 4 months) of starting ADT. Docetaxel will be given alone every three weeks until 6 total infusions of docetaxel are complete.

In all three arms, the first docetaxel infusion is given as an inpatient to help with the blood draws required for the study. After the first docetaxel, all other docetaxel treatments will be given as an outpatient in the day hospital unless there is a need to do it as an inpatient. The vaccine injections are given in the day hospital unless you admitted as an inpatient for any reason. If you are randomized to Arm B, the vaccine and docetaxel must be given at least 20-48 hours apart. You will need to return the following day to get the docetaxel infusion.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

For more information about the vaccine and the booster vaccines, please see below under Vaccinia Virus and Fowlpox Virus.

Once we know which group/arm you will join, we will provide you with a schedule. You can expect blood tests, vital signs and a physical exam with each clinic visit.

As part of this study, we will look for any signs that your cancer is getting worse:

- Your PSA level will be checked at each visit when blood is taken.
- Bone scan will be done at baseline and as needed based on your symptoms.
- CT scan of the chest, abdomen, and pelvis or MRI will be done at baseline and as needed based on your symptoms.

### Research blood samples

An important part of this study is testing the effects of this treatment on your tumor and immune system. Research tests will be done on blood taken at different times during the study. The NIH has set a limit on the maximum amount of blood that can be taken for research. This limit is based on your age. For adults, no more than 37 tablespoons can be taken over an 8-week period. All patients who join the study will have blood samples drawn for pharmacokinetic (PK) studies. PK studies try to find out how the body affects the drug after it has been given to a person. We will do this study with the first docetaxel treatment. We will collect the blood before you start your initial infusion of docetaxel, about 5 minutes before the docetaxel infusion ends, 15 minutes, 30 minutes, 3 hours, 6 hours, 12 hours and 24 hours after the end of the docetaxel infusion. We will need to admit you into the hospital to make it easier on you to collect the sample. We will insert two IV lines (one in each arm). One IV line is for the chemotherapy infusion, the other IV line is for the blood collection.

In addition, we may at various time points during the study, collect blood samples to study your immune system (group of cells and organs in the body that recognize and fight infection). The samples we collect will help us better understand how the vaccine works inside the human body. The samples are for research purposes only.

#### <u>Tumor biopsy (optional)</u>

We would like to collect tumor samples by doing biopsies at two time points during the study (before you begin treatment and after you receive 2 cycles of vaccine therapy). For patients in Arm C it will be before you start vaccine and after vaccine is completed its full course. These biopsies will help us evaluate immune changes within the tumor. The decision for a biopsy will be based on the level of risk. The biopsy procedure usually causes only brief discomfort at the site from which the biopsy is taken. Rarely, infection or bleeding may occur at the needle site.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| Study | MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|---|
|---|---|---|

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

A separate consent form will be provided to you at the time of the biopsy for you to grant permission to that procedure if you agree to the biopsy. You can participate in the study even if you decide not to undergo the biopsies.

## When you are finished taking the drugs (treatment)

When you stop chemotherapy and vaccine, we will ask you to return to our clinic for a safety visit about 3-5 weeks after your last treatment. During the safety visit we will collect blood samples, do vital signs and physical exam. We may ask you to do other tests and procedures that are part of regular cancer care, or have a CT scan of the chest, abdomen, and pelvis or MRI and bone scan if needed to evaluate your cancer. Please note, you will continue ADT indefinitely which is considered the standard of care for this type of prostate cancer.

After the safety visit, we will follow you at NIH every 12 weeks. During the follow up visits you will have blood tests (including PSA), vital signs and physical exam. When the cancer requires treatment again (disease progression) we will take you off this study and ask you to enroll on a long term follow up study for patients who receive vaccine injections. On the long term follow up study we will contact you once a year until death or until you refuse further follow up. We will ask you about your PSA and prostate cancer treatment. See the section below on *Gene Therapy Long Term Follow up* below for additional information.

### Gene Therapy Long Term Follow up

You will be followed on a separate protocol once you are off this study. The Food and Drug Administration (FDA) requires that people who receive gene therapy are watched even after they complete therapy. Once you have finished therapy, you will be watched for up to 15 years to see how well you are doing. At least, you will be asked to have a routine physical exam each year for five years following your last vaccination. You will be asked questions about your health such as whether you have developed any new cancers or problems with your blood or immune system (the organs and cells that defend your body against infections and other diseases). You will also be asked whether you have had a hospital stay for something you did not expect and the medicines you are taking. You will be called by telephone for more information about your health each year for 15 years following your last treatment. The FDA will have access to this information. For this reason, we ask that you continue to provide us with a current address and telephone number, even after you complete this research study.

Please note, this therapy involves two immune stimulating therapies that have shown no evidence thus far that they impact your genes/genetics.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study | MEDICAL RECORD |
|---|---|
|---|---|

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

## **Risks or Discomforts of Participation**

#### Vaccinia Virus

The first vaccine injection you will receive is PROSTVAC-Vaccinia. It is made from the vaccinia virus. Vaccinia virus has been given to hundreds of millions of people worldwide to prevent the disease smallpox.

A potential problem that can occur with vaccinia vaccination is the accidental spread of the virus to another part of your body. This happens rarely (incidence 1 in 4000 in some reports), however, it is very important to protect against it. You can transfer the virus to your eye and mucous membranes (inner lining) of the nose, mouth or genitals by scratching the vaccination site and then rubbing the eye or an open skin area. If you participate in this study, you will have to take special care of your vaccination site and wash your hands often to prevent spreading the virus.

You may "shed" live virus from the vaccination site until the vaccination site heals completely. Until the site has healed completely, you could spread the virus to others. You must avoid close contact with the following people for approximately 3 weeks after the vaccinia vaccination only:

- persons with weak immune systems such as persons with leukemia or lymphoma, people
  with AIDS, or those receiving treatment to lower their immune system (for example, after
  organ transplantation).
- persons with eczema or other skin disorders that leave the skin open like surgical wounds, burns, chicken pox, or skin injuries like deep cuts.
- pregnant or breast-feeding women
- or, children under 3 years of age

"Close contact" means that these people share your house with you, are in physical contact with you, come in contact with your bed linens or clothes, and/or you take care of them and touch them.

#### How is the vaccine given?

In clinical studies of PROSTVAC, the vaccine is given by injection under the skin (subcutaneous). A dressing will be placed over the vaccination site to reduce the risk of accidental spreading. It is very important that you keep the vaccination site covered. Hand washing is also necessary. A dressing is placed over the vaccination site and you will be given instructions on how to take care of it.

#### What other risks or side effects can I expect from the vaccinia vaccine?

Most patients may get some redness and swelling in the surrounding area, approximately 1-4 inches (2-10 centimeters) in size. This lasts for about 7-14 days and may be come with itching and soreness. There is typically full healing and no leftover scarring from the subcutaneous injection. On average, vaccinia stays active in your body for about 10-14 days. Before you receive your next vaccine, you will be evaluated for any signs of bacterial infection, blisters, vesicles, (lesions seen on your skin at or around your vaccine site) or signs of vaccinia infection.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

Possible side effects can also be related to allergic responses the vaccine itself. An allergic reaction to the study vaccine may be development of a rash or hives within 7 to 10 days after vaccination, which usually gets better within 2 to 4 days. Rarely, a serious allergic reaction requiring hospitalization may occur.

Serious side effects from the vaccinia vaccine are most common in young children, subjects with disorders of the immune system, and individuals with skin disorders. That is why precautions are taken to exclude such individuals from exposure.

Serious reactions such as post-vaccinia encephalomyelitis ("brain inflammation") can lead to coma and death. Growth of a large non-healing sore and death are the most severe complications after vaccination. They occur mostly in very young children who are exposed to vaccinia for the first time, or in people with weak immune system; these people are not eligible for this study and must be avoided after vaccination. The death rate for people receiving revaccination with vaccinia for smallpox is about 1 in 10 million.

These serious reactions have not been seen in any subjects treated with PROSTVAC-V to date.

If symptoms for any of the vaccinia complications listed above appear, or if close contact occurs between a vaccinia-vaccinated patient and another at risk person should happen, contact the protocol investigator or study coordinator right away. You will be given the contact information. There are ways to treat the exposure if caught early.

#### Fowlpox Virus

PROSTVAC-F (the second and later doses of PROSTVAC) is based on fowlpox virus. Fowlpox virus naturally infects birds, not mammals, and has been researched and used in other vaccines for at least twenty years. The virus does not grow (replicate) in human cells and is not known to cause human disease. Previous studies have shown that using the fowlpox-based vaccine after the vaccinia-based vaccine causes a better clinical response compared to using the virus alone or using fowlpox before vaccinia. The vaccines including fowlpox virus have been given in research studies to both animals and humans for HIV, malaria and cancer.

#### What risks or side effects can I expect from the fowlpox vaccine?

Side effects from fowlpox are mild and could include injection site reactions, fever, fatigue (feeling very tired), anemia (low red blood cell count) and leucopenia (low white blood cell count). With any experimental treatment, there is the risk of unexpected and serious or deadly complications even if they have not been seen previously.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

# Additional risks and side effects related to the vaccine therapy with PROSTVAC-V and PROSVTAC-F

#### Likely:

- Injection site reaction (pain, swelling, itching, induration, and redness)
- Tiredness (fatigue or lethargy), general or leg weakness
- Fever
- Shaking chills (feeling cold)
- Nausea
- Swollen glands that may become bigger and tender

#### Less likely:

- Headache
- Allergic reaction
- Sweating
- Wound problems
- Vomiting
- Confusion and disorientation (not knowing where you are)
- Loss of appetite
- Yeast infection
- Constipation
- Cough
- Diarrhea
- Indigestion
- Facial tingling or numbness
- Muscle ache
- Itching

#### Rare but serious:

• An uncommon blood condition called thrombotic thrombocytopenic purpura (TTP). One patient treated with this vaccine developed TTP. It is not known if this was related to the vaccine or from something else. TTP is a serious disease that is associated with low blood counts (both red blood cells that carry oxygen and platelets that help your blood clot), bleeding, fever, neurologic symptoms (such as changes in level of alertness including coma, headache, difficulty speaking, confusion or paralysis) and kidney problems. The symptoms are caused by clots that form or spread to other organs. This can usually be treated with a therapy. Should you go on this trial, we will follow you closely for any signs or symptoms of this disease.

#### Other Potential Side Effects

Additional side effects could be related to the immune response to the PSA and/or TRICOM proteins that are part of the vaccines. Some normal human cells (such as normal prostate cells) have these proteins on their surface. If the vaccine causes an immune reaction against these normal

| PATIENT IDENTIFICATION | <b>CONTINUATION SHEET for either:</b> |
|------------------------|---------------------------------------|
| | NIH-2514-1 (07-09) |
| | NIH-2514-2 (10-84) |
| | P.A.: 09-25-0099 |
| | File in Section 4: Protocol Consent |

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
| | Study |

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

cells, you could develop swelling or inflammation of these tissues. While unlikely, it is also possible that if you develop a very active antibody (immune) reaction after the vaccination, you could develop something called serum sickness which can cause fevers, rashes, joint pains, and less commonly, kidney failure and swelling of the blood vessels (vasculitis) or any part of your body. None of these symptoms have been observed to date in subjects receiving the Bavarian Nordic vaccines, but the possibility of their occurrence exists.

#### **Docetaxel Risks**

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Docetaxel, more than 20 and up to 100 may have:

- Swelling of the body
- Hair loss
- Change in nails
- Rash, itching
- Vomiting, diarrhea, nausea
- Sores in mouth which may cause difficulty swallowing
- Infection, especially when white blood cell count is low
- Anemia which may require blood transfusions
- Tiredness
- Numbness and tingling of the arms and legs
- Fever
- Swelling and redness of the arms, leg or face
- Pain
- Watering, itchy eyes

**CONTINUATION SHEET for either:** NIH 2514-1, Consent to Participate in A Clinical Research Study MEDICAL RECORD

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Docetaxel, more than 20 and up to 100 may have:

### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Docetaxel, from 4 to 20 may have:

- Severe skin rash with blisters and peeling which can involve inside of mouth and other parts of the body
- Belly pain
- Bruising, bleeding
- Liver damage which may cause yellowing of eyes and skin
- Kidney damage which may require dialysis
- Scarring of the lungs
- Blood clot which may cause swelling, pain, shortness of breath
- Abnormal heart rate
- Shortness of breath, wheezing
- Chest pain

#### RARE, AND SERIOUS

In 100 people receiving Docetaxel, 3 or fewer may have:

- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Liver damage which may cause yellowing of the eyes and skin

#### Risks to an Unborn Child and Sexual Partner

#### **Birth Control**

Your study doctor will discuss the risks to unborn children for drugs other than PROSTVAC that may be used in this study. The effects of PROSTVAC, if any, on unborn children are unknown. If your partner is capable of becoming pregnant and you wish to participate in this study, and you have not had your prostate or testicles removed, or you are not receiving continuous hormone therapy, then you must use a medically acceptable method of birth control and refrain from donating sperm while you are receiving study vaccine and for a period of at least 4 months after your last dose of study vaccine.

If your partner becomes pregnant during the course of treatment, you must inform your doctor immediately. Your doctor will ensure that you and your partner receive information about options

PATIENT IDENTIFICATION **CONTINUATION SHEET for either:** 

NIH-2514-1 (07-09)

NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

available to you in relation to pregnancy and that you and your partner are fully supported in whichever option you chose.

Acceptable birth control options for you and your partner include:

- surgical sterilization (you and/or your partner)
- approved hormonal contraceptives or therapies (such as birth control pills, Depo-Provera, or Lupron Depot)
- barrier methods (such as a condom or diaphragm) used with a spermicide
- an intrauterine device (IUD)

#### Other Risks

The study treatment may involve risks to you that are currently unknown. Your cancer may not get better or may become worse while you are in this study.

Risks from X-rays and / or Scans: Radiological testing, such as CT scans, MRIs, X-rays and/or radioactive drugs may be used to assess the treatment of your disease at various times during therapy. The cumulative radiation exposure from these tests is considered very small and is unlikely to adversely affect you or your disease. Because some of these tests require administration of contrast you could experience pain, bruising, and/or infection at the site of injection, or an allergic reaction to the contrast agent. Please notify the investigator if you know or suspect you are allergic to contrast dye.

ECG: There are no significant risks or discomforts associated with an ECG. Some patches will be adhered to your skin that may cause some reddening or slight itching.

Blood draws: There may be some side effects associated with the procedures for drawing blood in this study, but the person drawing your blood will attempt to minimize this discomfort. Side effects include pain and bruising in the area where the needle is inserted, lightheadedness, and rarely, fainting. When large amounts of blood are collected, low red blood cell count (anemia) is a risk.

#### **Potential Benefits of Participation**

#### Are there benefits to taking part in this study?

The aim of this study is to see if this PROSTVAC vaccine will cause your tumors to shrink. We do not know if you will receive personal medical benefit from taking part in this study. These potential benefits could include shrinking of your tumor or lessening of your symptoms, such as pain, that are caused by the cancer. Because there is not much information about the drug's

| PATIENT IDENTIFICATION | CONTINUATION SHEET for either: |
|------------------------|-------------------------------------|
| | NIH-2514-1 (07-09) |
| | NIH-2514-2 (10-84) |
| | P.A.: 09-25-0099 |
| | File in Section 4: Protocol Consent |

| MEDICAL RECORD | CONTINUATION SHEET for either:<br>NIH 2514-1, Consent to Participate in A Clinical Research Study<br>NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research<br>Study |
|---|---|
| | CONTENT TT MTCONT |

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

effect on your cancer, we do not know if you will benefit from taking part in this study, although the knowledge gained from this study may help others in the future who have cancer.

## **Alternative Approaches or Treatments**

#### What other choices do I have if I do not take part in this study?

Instead of being in this study, you have these options:

- Taking part in another study
- Getting treatment with standard therapy outside this study (ADT alone or ADT with chemotherapy)
- Observation only, where your doctor, depending on his clinical judgment and your opinion, follows your PSA and watches you for cancer recurrence.
- In June of 2017, new data indicated that an oral hormone therapy that is FDA approved for prostate cancer (abiraterone) can also be taken daily with ADT and improve survival compared to ADT alone. The best comparisons at this time suggest that this daily treatment may be equivalent to the 6 infusions of docetaxel chemotherapy.

Please talk to your doctor about these and other options.

### Research Subject's Rights

#### What are the costs of taking part in this study?

If you choose to take part in the study, the following will apply, in keeping with the NIH policy:

- You will receive study treatment at no charge to you. This may include surgery, medicines, laboratory testing, x-rays or scans done at the Clinical Center, National Institutes of Health (NIH), or arranged for you by the research team to be done outside the Clinical Center, NIH if the study related treatment is not available at the NIH.
- There are limited funds available to cover the cost of some tests and procedures performed outside the Clinical Center, NIH. You may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the Clinical Center, NIH.
- Once you have completed taking part in the study, medical care will no longer be provided by the Clinical Center, NIH.

| MEDICAL RECORD | CONTINUATION SHEET for either:<br>NIH 2514-1, Consent to Participate in A Clinical Research Study<br>NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research<br>Study |
|---|---|
| | CONTENT TT MTCONT |

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

## Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The National Cancer Institute (NCI) and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Cancer Institute Institutional Review Board
- The study Sponsor, Center for Cancer Research, or their agent(s)
- Qualified representatives from Bavarian Nordic, Inc., the pharmaceutical company who produces PROSTVAC vaccine.

A description of this clinical trial will be available on <a href="http://www.Clinicaltrials.gov">http://www.Clinicaltrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

#### **Certificate of Confidentiality**

To help us protect your privacy, we have obtained a Certificate of Confidentiality. The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

You should also know that there are several circumstances in which the Certificate does not provide coverage. These include when information:

- will be used for auditing or program evaluation internally by the NIH; or
- must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA).
- is necessary for your medical treatment and you have consented to this disclosure;
- is for other research.

In addition, identifiable, sensitive information protected by this Certificate cannot be admissible as evidence or used for any purpose in any action, suit, or proceeding without your consent.

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

| Study | MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|---|
|---|---|---|

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

The Certificate of Confidentiality will not protect against the required reporting by hospital staff of information on suspected child abuse, reportable communicable diseases, and/or possible threat of harm to self or others.

## **Stopping Therapy**

You will continue to receive therapy and medical follow-up until:

- The study is completed;
- You decide that you no longer wish to participate in the study;
- You experience unacceptable side effects;
- Your cancer gets worse;
- You need to start another kind of therapy (called androgen deprivation therapy) for your cancer
- The doctor feels that it is unsafe for you to continue;
- New information becomes available that suggests another treatment would be better for you; or
- The study is stopped.

You can stop taking part in the study at any time. However, if you are thinking about dropping out of the study, please tell your research team so they can tell you how to end your participation safely.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to Bavarian Nordic, Inc. or designated representatives. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases cannot be recalled and destroyed.

#### **Conflict of Interest**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a Protocol Review Guide. You may ask your research team for a copy of the Protocol Review Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines but they do not need to report their personal finances to the NIH.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

Members of the research team working on this study may have up to \$15,000 of stock in the companies that make products used in this study. This is allowed under federal rules and is not a conflict of interest.

The National Institutes of Health and the research team for this study are using vaccine developed in collaboration with the National Cancer Institute under a Cooperative Research and Development Agreement with Bavarian Nordic, Inc. The company also provides financial support for this study.

#### Use of Specimens and Data for Future Research

To advance science, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the information must apply to the database and be approved. Researchers use specimens and data stored in scientific databases to advance science and learn about health and disease.

We plan to keep some of your specimens and data that we collect and use them for future research and share them with other researchers. We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. Your specimens and data will be used for research purposes only and will not benefit you. It is also possible that the stored specimens and data may never be used. Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

If you do not want your stored specimens and data used for future research, please contact us in writing and let us know that you do not want us to use your specimens and/or data. Then any specimens that have not already been used or shared will be destroyed and your data will not be used for future research. However, it may not be possible to withdraw or delete materials or data once they have been shared with other researchers.

#### **Optional Imaging**

Another way to monitor your tumor for any signs that your cancer is recurring or getting worse is with an endorectal MRI (an MRI image taken from inside the rectum) and Sodium Fluoride (NaF) PET scans. These scans will be done at baseline and, every 12 months until progression or and then at progression.

These scans to be performed are exclusively for research purposes and will not benefit you. It might help other people in the future. Even if you decide to have the scans you can change your mind at any time. The decision to participate in this part of the research is optional, and no matter what you decide to do, it will not affect your care.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either:<br>NIH 2514-1, Consent to Participate in A Clinical Research Study<br>NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research<br>Study |
|---|---|

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

You will be given the opportunity to decide whether you want to participate at the time of the procedure.

#### Research Radiation Risks:

This research study may involve exposure to radiation from a low dose CT with NaF PET scan at baseline and every 12 months until progression or at progression. This radiation exposure is not required for your medical care and is for research purposes only. From participating in this, the total amount of radiation you will receive is 1.2 rem which is below the guideline of 5.0 rem per year allowed for research subjects by the NIH Radiation Safety Committee. The average person in the United States receives a radiation exposure of 0.3 rem per year from natural sources, such as the sun, outer space, and the earth's air and soil. If you would like more information about radiation, please ask the investigator for a copy of the pamphlet, <u>An Introduction to Radiation for NIH Research Subjects</u>.

While there is no direct evidence that the amount of exposure received from participating in this study is harmful, there is indirect evidence it may not be completely safe. There may be a very slight increase in the risk of cancer.

Please tell your doctor if you have had any radiation exposure in the past year, either from other research studies or from medical tests or care, so we can make sure that you will not receive too much radiation. Radiation exposure includes x-rays taken in radiology departments, cardiac catheterization, and fluoroscopy as well as nuclear medicine scans in which radioactive materials were injected into your body.

MEDICAL RECORD

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

STUDY NUMBER: 16-C-0048

CONTINUATION:  pages

#### OTHER PERTINENT INFORMATION

1. Confidentiality. When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

The Federal Privacy Act protects the confidentiality of your NIH medical records. However, you should know that the Act allows release of some information from your medical record without your permission, for example, if it is required by the Food and Drug Administration (FDA), members of Congress, law enforcement officials, or authorized hospital accreditation organizations.

- 2. Policy Regarding Research-Related Injuries. The Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the National Institutes of Health, the Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.
- 3. Payments. The amount of payment to research volunteers is guided by the National Institutes of Health policies. In general, patients are not paid for taking part in research studies at the National Institutes of Health. Reimbursement of travel and subsistence will be offered consistent with NIH guidelines.
- **4. Problems or Questions.** If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Ravi Madan, M.D., Building 10, Room 13N240, Telephone: 301-480-7168. You may also call the Clinical Center Patient Representative at 301-496-2626. If you have any questions about the use of your specimens or data for future research studies, you may also contact the Office of the Clinical Director, Telephone: 240-760-6070.
- **5. Consent Document.** Please keep a copy of this document in case you want to read it again.

PATIENT IDENTIFICATION

**CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)** 

• Adult Patient or NIH-2514-1 (07-09) · Parent, for Minor Patient

P.A.: 09-25-0099

MEDICAL RECORD

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

STUDY NUMBER: 16-C-0048 CONTINUATION:  pages

| COMPLETE APPROPRIATE ITEM(S) BELOW: | | | |
|---|---|---|---|
| A. Adult Patient's Consent | | B. Parent's Permission for Minor Patient. | |
| I have read the explanation about this study<br>and have been given the opportunity to<br>discuss it and to ask questions. I hereby<br>consent to take part in this study. | | I have read the explanation about this study<br>and have been given the opportunity to<br>discuss it and to ask questions. I hereby give<br>permission for my child to take part in this<br>study. | |
| | | (Attach NIH 2514-2, Minor's As applicable.) | sent, if |
| Signature of Adult Patient/<br>Legal Representative | Date | Signature of Parent(s)/ Guardian | Date |
| Print Name | | Print Name | |
| C. Child's Verbal Assent (If Ap | plicable) | | |
| The information in the above consparticipate in the study. | ent was desc | ribed to my child and my child agi | rees to |
| Signature of Parent(s)/Guardian | Date | Print Name | |
| THIS CONSENT DOCUMENT HAS BEEN APPROVED FOR USE FROM OCTOBER 15, 2020 THROUGH OCTOBER 14, 2021. | | | |
| Signature of Investigator | Date | Signature of Witness | Date |
| Print Name | | Print Name | |

PATIENT IDENTIFICATION

# **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)**

• Adult Patient or NIH-2514-1 (07-09)

• Parent, for Minor Patient

P.A.: 09-25-0099